CLINICAL TRIAL: NCT01630408
Title: A Pilot Study of the Effects of Active VItamin D on Left Atrial Volume Index in Patients With Heart Failure and Preserved Ejection Fraction
Brief Title: The Effects of Active VItamin D on Left Atrial Volume Index
Acronym: AVID-LAVI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator decided not to pursue.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ravi Thadhani, Director of Clinical Research in Nephrology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVID-LAVI
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Last update posted 2013-08-16 (Estimated); Status verified 2013-08

CONDITIONS: Heart Failure
Keywords: Preserved ejection fraction; Left ventricular hypertrophy; Activated vitamin D; Cardiac lusitropic effect; Hospitalizations
MeSH Terms: conditions — Heart Failure; Hypertrophy, Left Ventricular | interventions — paricalcitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paricalcitol (Experimental): Paricalcitol oral capsules (1 mcg per day for 48 weeks)
  Interventions: Drug: Paricalcitol

INTERVENTIONS:
Drug: Paricalcitol — Paricalcitol oral capsules 1 mcg/day for 48 weeks
  Other Names: Zemplar®

SUMMARY:
This is a pilot feasibility study to determine the effects of an activated vitamin D compound (paricalcitol) on heart structure (size) and function (ability to relax) in patients with normal kidney function and a form of heart failure known as HFPEF (heart failure and preserved ejection fraction). This study will also examine heart failure-related hospitalizations and changes in cardiac-stretch and biological markers that are believed to change along with heart size. Patients in this pilot study will be treated for a period of 48 weeks with paricalcitol at a dose previously approved by FDA (1 mcg per day) and followed-up for 4 weeks after treatment is completed.

DETAILED DESCRIPTION:
Heart failure (HF) is among the top ten causes of hospitalizations in the US. It is estimated that ~40-50% of patients with HF have preserved ejection fraction (EF). Patients with heart failure and preserved ejection fraction (HFPEF) have normal systolic function, but impaired cardiac relaxation. The main causes of HFPEF include left-ventricular hypertrophy (LVH) and hypertension, hypertrophic cardiomyopathy, aortic stenosis with a normal EF, coronary artery disease and restrictive cardiomyopathies.

Only a few small clinical trials have tested therapeutic interventions in patients with HFPEF, producing either small or negative effects. Relatively few drugs have effects on cardiac relaxation and are not candidates for chronic use, as they may have significant side effect profiles and/or are inconvenient to administer. Paricalcitol, an FDA-approved activated form of vitamin D, has been shown to slow LVH progression and improve parameters associated with diastolic function in animal models (see refs). Treatment with paricalcitol has also been associated with decreased cardiovascular morbidity and mortality in a historical cohort study of patients with end-stage renal disease (see refs).

This is a single-center, single-arm, pilot study in 20 patients with HFPEF and normal renal function on stable medical therapy to evaluate the effects of paricalcitol on cardiac structure and function.

ELIGIBILITY:
Inclusion Criteria:

* Sign informed consent.
* Willing and able to adhere to all study-related procedures, including study medication regimen.
* ≥ 18 years old.
* Previous clinical diagnosis of heart failure with preserved ejection fraction: NYHA Class II-IV.
* Satisfy these echocardiographic criteria within the last year: Left ventricular ejection fraction ≥ 50%, cardiac magnetic resonance or ventriculogram; Left atrial size ≥ 4 cm in long axis or > 5.2 cm in four chamber length; Septal wall thickness > 1.2 cm (females) or 1.3 cm (males); Doppler evidence of moderate or severe diastolic dysfunction (≥ Grade II) by transmitral inflow, pulmonary venous flow, color M-mode and/or tissue Doppler (per European Society of Cardiology guidelines).
* Experienced ≥ 1 of the following in last 12 months: Hospitalization for acute heart failure (primary diagnosis); Long term treatment with loop diuretic; Mean pulmonary capillary wedge pressure ≥ 16 mm Hg at catheterization for dyspnea; Left ventricular end diastolic pressure (LVEDP) ≥ 19 mm Hg at catheterization for dyspnea; Acute treatment with intravenous loop diuretic or hemofiltration.
* On stable medical therapy in last 30 days before study entry (defined as no change in angiotensin converting enzyme inhibitors [ACEI], angiotensin receptor blockers, aldosterone inhibitors, beta-blockers or calcium channel blockers.
* Satisfy these criteria at initial lab screening: Estimated glomerular filtration rate (eGFR) ≥ 30 ml/min; Corrected serum Ca 8.0-10.0 mg/dL (2.0-2.5 mmol/L); Phos ≤ 5.2 mg/dL (1.68 mmol/L); Serum albumin ≥ 3.0 g/dL (30 g/L);
* Negative serum pregnancy test for females of childbearing potential (within 2 weeks of starting study treatment).
* Women of childbearing potential must be practicing barrier/oral contraception during study-related treatment, or be surgically sterile or one year post-menopausal, be non-nursing and non-pregnant.

Exclusion Criteria:

* Taking > 1,000 IU of vitamin D preparation daily within last 30 days.
* Received activated vitamin D preparation including paricalcitol (Zemplar®), doxercalciferol (Hectorol®) or calcitriol (Rocalctrol®, Calcijex®) within last 90 days prior to study entry.
* History of nephrolithiasis.
* Poorly controlled hypertension (systolic blood pressure > 180 mmHg and/or diastolic blood pressure > 110 mmHg at Screening; confirmed by repeat).
* Secondary hypertension (i.e. renal artery stenosis, primary aldosteronism or pheochromocytoma).
* Severe hepatic impairment.
* Use of known inhibitors (ie, ketoconazole) or inducers (ie, carbamazepine) of cytochrome P450 3A (CYP3A) within 2 weeks prior to taking study drug.
* HIV positive.
* Condition with prognosis < 1 year at study entry other than heart failure.
* Significant valvular disease defined as moderate or severe aortic or mitral stenosis, mitral or aortic regurgitation.
* Infiltrative cardiac disease (sarcoid, amyloid, hemochromatosis, lymphoma, etc.).
* Arrhythmogenic right ventricular cardiomyopathy.
* Active myocarditis.
* Constrictive or restrictive pericarditis.
* Acute coronary artery disease symptoms defined as emergency department visit or hospital admission with unstable angina, ST-elevation myocardial infarction (STEMI), non-ST-elevation myocardial infarction (NSTEMI), percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG) within 90 days before study entry.
* Poor echocardiographic windows.
* Current active treatment in another investigational study or participation in another investigational study within 1 month before screening.
* Active malignancies except in situ carcinoma of the cervix, localized squamous or basal cell carcinoma of skin.
* Other serious concurrent or recent medical or psychiatric condition which, in Investigator's opinion, makes the patient unsuitable for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2014-05 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Change in left atrial volume index (LAVI) by transthoracic echocardiography. | Baseline and Week 48
  The analysis will include all patients with at least two echocardiographic studies (baseline and one follow up). The primary endpoint will be determined upon completion of the study (ie, when all enrolled patients have been treated for up to 48 weeks with study medication).

SECONDARY OUTCOMES:
Number of and time-to-first heart failure-related hospitalizations | 52 weeks
Overall cardiac and non-cardiac mortality rates | 52 weeks
Changes in biological, inflammatory, LVH and strain biomarkers that have been linked to cardiovascular disease. | Baseline and 48 weeks
  High-sensitivity troponin-T, NT-proBNP, high-sensitivity C-reactive protein, propeptide procollagen type I, ST-2, Galectin-3, GDF-15 and osteoprotegerin
Changes in standard mineral metabolite parameters (calcium, phosphorus, calcium-phosphate-product and PTH) | Baseline and 48 weeks
Changes in self-reported Patient Global Assessment | Baseline and 48 weeks
Change in diastolic function parameters (including E, A, IVRT, DT) | Baseline and Week 48
Change in tissue doppler parameters (including Ea, Aa) | Baseline and Week 48
Change in pulmonary venous inflow (including S, D, a reversal) | Baseline to Week 48
Change in cardiac ejection fraction | Baseline and Week 48
Change in end-diastolic and end-systolic left ventricular internal dimension | Baseline and Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Hector Tamez, MD, MPH, Principal Investigator — Massachusetts General Hospital; Ravi Thadhani, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Bodyak N, Ayus JC, Achinger S, Shivalingappa V, Ke Q, Chen YS, Rigor DL, Stillman I, Tamez H, Kroeger PE, Wu-Wong RR, Karumanchi SA, Thadhani R, Kang PM. Activated vitamin D attenuates left ventricular abnormalities induced by dietary sodium in Dahl salt-sensitive animals. Proc Natl Acad Sci U S A. 2007 Oct 23;104(43):16810-5. doi: 10.1073/pnas.0611202104. Epub 2007 Oct 17. PMID 17942703
- [Background] Wu J, Garami M, Cheng T, Gardner DG. 1,25(OH)2 vitamin D3, and retinoic acid antagonize endothelin-stimulated hypertrophy of neonatal rat cardiac myocytes. J Clin Invest. 1996 Apr 1;97(7):1577-88. doi: 10.1172/JCI118582. PMID 8601621
- [Background] Weishaar RE, Simpson RU. Vitamin D3 and cardiovascular function in rats. J Clin Invest. 1987 Jun;79(6):1706-12. doi: 10.1172/JCI113010. PMID 3034981
- [Background] Teng M, Wolf M, Lowrie E, Ofsthun N, Lazarus JM, Thadhani R. Survival of patients undergoing hemodialysis with paricalcitol or calcitriol therapy. N Engl J Med. 2003 Jul 31;349(5):446-56. doi: 10.1056/NEJMoa022536. PMID 12890843